CLINICAL TRIAL: NCT05054725
Title: A Phase 2, Open-Label, Multicenter Study of the Combination of RMC-4630 and Sotorasib for Non-Small Cell Lung Cancer Subjects With KRASG12C Mutation After Failure of Prior Standard Therapies
Brief Title: Combination Study of RMC-4630 and Sotorasib for NSCLC Subjects With KRASG12C Mutation After Failure of Prior Standard Therapies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revolution Medicines, Inc. (Industry)
Collaborators: Sanofi (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RMC-4630-03
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: SHP2; NSCLC; KRAS G12C; BRAF Class 1/2/unclassified; KRAS amplification; KRAS mutation; STK11/LKB1; KEAP1; PIK3CA; ATRX; BRCA2; carcinoma, non-small lung cancer; bronchial neoplasms; lung neoplasms; respiratory tract neoplasms; neoplasms by site; neoplasms; lung diseases; respiratory tract diseases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Hereditary Sensory and Autonomic Neuropathies; Carcinoma; Bronchial Neoplasms; Lung Neoplasms; Respiratory Tract Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases | interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RMC-4630 and sotorasib, Safety Run-in (Experimental): Safety Run-In:
  RMC-4630 and sotorasib
  Interventions: Drug: RMC-4630; Drug: Sotorasib
- RMC-4630 and sotorasib, Expansion (Experimental): Dose Expansion:
  RMC-4630 and sotorasib
  Interventions: Drug: RMC-4630; Drug: Sotorasib

INTERVENTIONS:
Drug: RMC-4630 — RMC-4630 administered orally as a capsule
  Other Names: SAR442720
Drug: Sotorasib — Sotorasib administered orally as a tablet
  Other Names: AMG 510; Lumakras

SUMMARY:
The purpose of this study is to evaluate the antitumor effects of sotorasib and RMC-4630 in subjects with KRASG12C mutant NSCLC

DETAILED DESCRIPTION:
This is a phase 2 multicenter, open-label study evaluating the efficacy, safety, tolerability, and pharmacokinetics (PK) of RMC-4630 in combination with sotorasib in subjects with KRASG12C mutant NSCLC after failure of prior standard therapies.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥18 years of age.
* Subject must have pathologically documented, locally advanced or metastatic KRASG12C NSCLC (not amenable to curative surgery) that has progressed on prior standard therapies (no more than 3 prior lines of therapies are allowed)

Exclusion Criteria

* Primary central nervous system (CNS) tumors
* Known or suspected leptomeningeal or brain metastases or spinal cord compression
* Clinically significant cardiac disease
* Known impairment of GI function that would alter the absorption
* Active autoimmune disease requiring systemic treatment within past 2 years
* History of severe allergic reactions to any of the study intervention components
* Major surgical procedures within 28 days or non-study-related minor procedures within 7 days of treatment.
* Prior therapy with KRASG12C inhibitor and/or SHP2 inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Revolution Medicines, Inc., Study Director — Revolution Medicines, Inc.
Locations (60):
- United States (23):
  - Florida Cancer Specialists, Fort Myers, Florida
  - BRCR Medical Center Inc., Plantation, Florida
  - Cancer Specialists of North Florida, Saint Augustine, Florida
  - GenHarp Clinical Solutions, Evergreen Park, Illinois
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - New England Cancer Specialists, Scarborough, Maine
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New Jersey Center for Cancer Research, Brick, New Jersey
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Roswell Park cancer Institute, Buffalo, New York
  - Clinical Research Alliance, Inc., New York, New York
  - Zangmeister Cancer Center, Columbus, Ohio
  - Charleston Oncology, Charleston, South Carolina
  - Tennessee Oncology, Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - CHRISTUS St. Michael-Colom and Carney Clinic P.A, Texarkana, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer specialists, P.C., Vancouver, Washington
- Australia (3):
  - South West Oncology, Warrnambool, Victoria
  - Blacktown Hospital, Blacktown
  - Goulburn Valley Health, Shepparton
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - William Osler Health System, Mississauga, Ontario
- France (2):
  - APHM Hopital Nord, Service d'Oncologie Multidisciplinaire et innovations therapeutics, Marseille
  - Hospital Larrey Universite Paul Sabatier, Toulouse
- Germany (10):
  - Klinikum Esslingen GmbH, Esslingen am Neckar, Baden-Wurttemberg
  - Asklepios Fachkliniken Munchen, Gauting, Bavaria
  - Lungenklinik Hemer, Hemer, North Rhine-Westphalia
  - Bethanien Hospital Moers, Moers, North Rhine-Westphalia
  - Comprehensive Cancer Center Mainfranken, University Wuerzburg, Homburg, Saarland
  - Lung Cancer Center, University of Saarland, Homburg, Saarland
  - POIS Sachsen GmbH, Leipzig, Saxony
  - Charite Benjamin Franklin Comprehensive Cancer center, Berlin
  - Evangelische Lung Clinic, Berlin
  - Hamato-Onkologie Hamburg, Hamburg
- Italy (3):
  - Azienda Ospedaliera dei Colli, Napoli, Campania
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Orbassano, Piedmont
  - Istituto Europeo Di Oncologia, Milan
- South Korea (4):
  - Chungbuk National University Hospital, Cheongju-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Complejo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario y Politecnico La Fe, Valencia
- Taiwan (5):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - E-DA Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This Phase 2 study (RMC-4630-03) had a safety run-in period in which RMC-4630 was administered at 140 mg twice weekly (BIW) on D1D2 of each week in a 21-day cycle and sotorasib 960 mg once daily (QD) in a 21-day cycle as the starting dose with the option of escalating to RMC-4630 200 mg BIW on D1D2 of each week in a 21-day cycle. Patients were evaluated for dose limiting toxicities (DLTs).
Groups:
- RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD; RMC-4630 200 mg D1D2 + Sotorasib 960 mg QD: The two arms have been broken down per dose level rather than by phase or cohort per the CSR, which is provided to FDA and not uploaded to ct.gov. Participants were administered 140 or 200 mg of RMC-4630 twice weekly (BIW) on D1D2 of each week in a 21-day cycle and Sotorasib 960 mg once daily (QD) in a 21-day cycle. The 140mg and 200mg dose levels were explored at the safety run-in stage, and after completion of the safety run-in (DLT clearance) of both dose levels, additional patients were enrolled at both dose levels for the purpose of dose optimization before selecting the final expansion dose. Therefore, both the 140mg and 200mg dose levels included patients in the safety-run in and dose optimization. After that, 200mg was identified as the RP2D dose, which moved to the expansion phase.
  Statistical analysis for all sections in the results was performed for all treated patients by dose level, i.e., 140mg vs 200mg. For patients enrolled at the RP2D dose level of 200mg, analysis was further performed based on mutation status, i.e., cohorts 1 vs 2.
Period: Overall Study
Arm/Group | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD | RMC-4630 200 mg D1D2 + Sotorasib 960 mg QD
Started | 4 | 43
Completed | 0 | 3
Not Completed | 4 | 40
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Sponsor's Decision to Terminate the Study | 0 | 3
Not completed — Death | 1 | 21
Not completed — Sponsor amended protocol to terminate Long Term Follow Up (LTFU) | 0 | 3
Not completed — PI's decision that there is no benefit from LTFU | 0 | 6
Not completed — Due to AE#17 - Angiosarcoma of the breast with possible relation to study drug | 0 | 1
Not completed — Agreed between patient and PI as safety follow up is not for benefit of the patient | 0 | 1
Not completed — Physician discretion due to subject progression | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD | RMC-4630 200 mg D1D2 + Sotorasib 960 mg QD | Total
Number analyzed (Participants) | 4 | 43 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 23 | 24
  >=65 years | 3 | 20 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 25 | 27
  Male | 2 | 18 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 1 | 8 | 9
  Race: Black or African American | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: White | 3 | 31 | 34
  Race: Other | 0 | 0 | 0
  Ethnicity: Hispanic or Latino | 0 | 2 | 2
  Ethnicity: Not Hispanic or Latino | 4 | 40 | 44
  Ethnicity: Missing/Not Reported | 0 | 1 | 1
  Race: Missing/Not Reported | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Assessed Per RECIST v1.1
Description: Evaluation of the antitumor effects of RMC-4630 and sotorasib in locally advanced or metastatic NSCLC patients with KRASG12C mutation with and without co-existing genetic aberrations in specific genes such as STK11/LKB1, KEAP1, and PIK3CA after failure of prior standard therapy. Objective Response Rate (%) is defined as the proportion of patients with Best Overall Response of confirmed CR, or PR. Response was confirmed by a repeat assessment no less than 28 days.
Time Frame: 31 months
Population: Objective Response Rate (%) is defined as the proportion of patients with Best Overall Response of confirmed CR, or PR.
Measure: Count of Participants; unit: Participants
Groups:
- RMC-4630 200 mg BIW D1D2 + Sotorasib 960 mg QD: The two arms have been broken down per dose level rather than by phase or cohort per the CSR, which is provided to FDA and not uploaded to ct.gov. Participants were administered 140 or 200 mg of RMC-4630 twice weekly (BIW) on D1D2 of each week in a 21-day cycle and Sotorasib 960 mg once daily (QD) in a 21-day cycle. The 140mg and 200mg dose levels were explored at the safety run-in stage, and after completion of the safety run-in (DLT clearance) of both dose levels, additional patients were enrolled at both dose levels for the purpose of dose optimization before selecting the final expansion dose. Therefore, both the 140mg and 200mg dose levels included patients in the safety-run in and dose optimization. After that, 200mg was identified as the RP2D dose, which moved to the expansion phase.
  Statistical analysis for all sections in the results was performed for all treated patients by dose level, i.e., 140mg vs 200mg. For patients enrolled at the RP2D dose level of 200mg, analysis was further performed based on mutation status, i.e., cohorts 1 vs 2.
Arm/Group | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD | RMC-4630 200 mg BIW D1D2 + Sotorasib 960 mg QD
Number analyzed (Participants) | 4 | 43
Participants | 0 | 11

2. Secondary Outcome: Clinically Significant Changes in Vital Signs
Description: Characterization of the safety, tolerability of RMC-4630 in combination with sotorasib for subjects with KRASG12C mutant NSCLC after failure of prior standard therapy
Time Frame: 31 months
Measure: Count of Participants; unit: Participants
Groups:
- RMC-4630 200 mg BIW D1D2 and Sotorasib 960 mg QD Safety-Run in, Optimization, Expansion: The two arms have been broken down per dose level rather than by phase or cohort per the CSR, which is provided to FDA and not uploaded to ct.gov. Participants were administered 140 or 200 mg of RMC-4630 twice weekly (BIW) on D1D2 of each week in a 21-day cycle and Sotorasib 960 mg once daily (QD) in a 21-day cycle. The 140mg and 200mg dose levels were explored at the safety run-in stage, and after completion of the safety run-in (DLT clearance) of both dose levels, additional patients were enrolled at both dose levels for the purpose of dose optimization before selecting the final expansion dose. Therefore, both the 140mg and 200mg dose levels included patients in the safety-run in and dose optimization. After that, 200mg was identified as the RP2D dose, which moved to the expansion phase.
  Statistical analysis for all sections in the results was performed for all treated patients by dose level, i.e., 140mg vs 200mg. For patients enrolled at the RP2D dose level of 200mg, analysis was further performed based on mutation status, i.e., cohorts 1 vs 2.
Arm/Group | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD | RMC-4630 200 mg BIW D1D2 and Sotorasib 960 mg QD Safety-Run in, Optimization, Expansion
Number analyzed (Participants) | 4 | 43
Participants | 0 | 0

3. Secondary Outcome: Clinically Significant Changes in Laboratory Tests
Description: as for outcome 2
Time Frame: 31 months
Measure: Count of Participants; unit: Participants
Arm/Group | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD | RMC-4630 200 mg D1D2 + Sotorasib 960 mg QD
Number analyzed (Participants) | 4 | 43
Participants
  Grade 3 Alanine Aminotransferase Increased | 1 | 5
  Grade 3 Aspartate Aminotransferase Increased | 2 | 5
  Grade 3 Bilirubin Increased | 0 | 5
  Grade 4 Alanine Aminotransferase Increased | 0 | 2
  Grade 4 Aspartate Aminotransferase Increased | 0 | 2

4. Secondary Outcome: Clinically Significant Changes in ECGs
Description: as for outcome 2
Time Frame: 31 months
Measure: Count of Participants; unit: Participants
Arm/Group | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD | RMC-4630 200 mg D1D2 + Sotorasib 960 mg QD
Number analyzed (Participants) | 4 | 43
Participants | 0 | 0

5. Secondary Outcome: Trough and Approximate Peak Concentrations of RMC-4630
Description: Characterization of PK of RMC-4630 in combination with sotorasib for subjects with KRASG12C mutant NSCLC.
Time Frame: 31 months
Population: Summary of PK of RMC-4630 concentration for subjects with KRASG12C mutant NSCLC (All Treated Subjects). Timepoints beyond Cycle 4 do not any value for the PK profile per sponsor. The decreasing number in participants analyzed is due to various factors such as missed samples or patient drop out as timepoints progressed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD | RMC-4630 200 mg D1D2 + Sotorasib 960 mg QD
Number analyzed (Participants) | 4 | 43
ng/ml
  Cycle 1 Day 15 pre-dose (within 1 hour pre-dose): number analyzed (Participants) | 4 | 33
  Cycle 1 Day 15 pre-dose (within 1 hour pre-dose) | 21.04 (138.51) | 27.55 (127.22)
  Cycle 1 Day 15 post-dose (2 hour +/- 10 minutes post-dose): number analyzed (Participants) | 4 | 33
  Cycle 1 Day 15 post-dose (2 hour +/- 10 minutes post-dose) | 187.64 (106.19) | 276.29 (122.66)
  Cycle 2 Day 1 pre-dose (within 1 hour pre-dose): number analyzed (Participants) | 4 | 32
  Cycle 2 Day 1 pre-dose (within 1 hour pre-dose) | 24.75 (269.94) | 22.34 (179.87)
  Cycle 3 Day 1 pre-dose (within 1 hour pre-dose): number analyzed (Participants) | 3 | 26
  Cycle 3 Day 1 pre-dose (within 1 hour pre-dose) | 82.40 (166.30) | 18.35 (155.47)
  Cycle 4 Day 1 pre-dose (within 1 hour pre-dose): number analyzed (Participants) | 3 | 24
  Cycle 4 Day 1 pre-dose (within 1 hour pre-dose) | 33.48 (535.67) | 14.67 (128.88)

6. Secondary Outcome: Trough and Approximate Peak Concentrations of Sotorasib
Description: Characterization of PK of RMC-4630 in combination with Sotorasib for subjects with KRASG12C mutant NSCLC
Time Frame: 31 months
Population: Summary of PK of Sotorasib concentration for subjects with KRASG12C mutant NSCLC (All Treated Subjects). Timepoints beyond Cycle 4 do not any value for the PK profile per sponsor. The decreasing number in participants analyzed is due to various factors such as missed samples or patient drop out as timepoints progressed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD | RMC-4630 200 mg D1D2 + Sotorasib 960 mg QD
Number analyzed (Participants) | 4 | 43
ng/mL
  Cycle 1 Day 15 pre-dose (within 1 hour pre-dose): number analyzed (Participants) | 4 | 34
  Cycle 1 Day 15 pre-dose (within 1 hour pre-dose) | 615.6 (173.5) | 375.4 (134.4)
  Cycle 1 Day 15 post-dose (2 hour +/- 10 minutes post-dose): number analyzed (Participants) | 4 | 33
  Cycle 1 Day 15 post-dose (2 hour +/- 10 minutes post-dose) | 6009.3 (119.2) | 4603.3 (77.3)
  Cycle 2 Day 1 pre-dose (within 1 hour pre-dose): number analyzed (Participants) | 4 | 31
  Cycle 2 Day 1 pre-dose (within 1 hour pre-dose) | 674.7 (193.2) | 336.4 (170.8)
  Cycle 3 Day 1 pre-dose (within 1 hour pre-dose): number analyzed (Participants) | 3 | 21
  Cycle 3 Day 1 pre-dose (within 1 hour pre-dose) | 342.2 (12146.3) | 190.3 (125.7)
  Cycle 4 Day 1 pre-dose (within 1 hour pre-dose): number analyzed (Participants) | 3 | 19
  Cycle 4 Day 1 pre-dose (within 1 hour pre-dose) | 803.5 (152.3) | 404.5 (367.3)

7. Secondary Outcome: Duration of Response (DOR) as Assessed Per RECIST v1.1
Description: Characterization of efficacy or RMC-4630 in combination with Sotorasib as assessed by DOR, DCR, PFS, and OS in patients with KRAS G12C-mutant locally advanced or metastatic NSCLC after failure of prior standard therapy
Time Frame: 31 months
Population: Duration of Response (DOR) Based on Investigator Assessments (Subjects with Confirmed CR or PR Responders only).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD | RMC-4630 200 mg BIW D1D2 + Sotorasib 960 mg QD
Number analyzed (Participants) | 0 | 11
months |  | 12.19 [8.31 to NA] — NE means 'The upper limit of the confidence interval is not estimable because not enough events occurred beyond that point.' For the NE, it means not applicable since there's no patient.

8. Secondary Outcome: Disease Control Rate (DCR) as Assessed Per RECIST v.1.1
Description: as for outcome 7
Time Frame: 31 months
Population: Disease Control Rate (%) is defined as the proportion of subjects with best overall response of CR, PR, or stable disease
Measure: Count of Participants; unit: Participants
Arm/Group | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD | RMC-4630 200 mg BIW D1D2 + Sotorasib 960 mg QD
Number analyzed (Participants) | 4 | 42
Participants | 3 | 34

9. Secondary Outcome: Progression-free Survival (PFS) as Assessed Per RECIST v1.1
Description: as for outcome 7
Time Frame: 31 months
Population: Summary of Progression-Free Survival (PFS) Based on Investigator Assessments (All Treated Subjects).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD | RMC-4630 200 mg BIW D1D2 + Sotorasib 960 mg QD
Number analyzed (Participants) | 4 | 43
months | 2.64 [1.28 to NA] — NE means 'The upper limit of the confidence interval is not estimable because not enough events occurred beyond that point.' For the NE, it means not applicable since there's no patient. | 7.66 [3.98 to 10.45]

10. Secondary Outcome: Overall Survival (OS)
Description: as for outcome 7
Time Frame: 31 months
Population: Summary of Overall Survival (OS) (All Treated Subjects).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD | RMC-4630 200 mg BIW D1D2 + Sotorasib 960 mg QD
Number analyzed (Participants) | 4 | 43
months | 5.80 [4.34 to NA] — NE means 'The upper limit of the confidence interval is not estimable because not enough events occurred beyond that point.' For the NE, it means not applicable since there's no patient. | 12.45 [9.72 to NA] — NE means 'The upper limit of the confidence interval is not estimable because not enough events occurred beyond that point.' For the NE, it means not applicable since there's no patient.

11. Secondary Outcome: Incidence, Nature and Severity of TEAEs, SAEs
Description: Characterization of the safety, tolerability of RMC-4630 in combination with sotorasib for patients with KRASG12C-mutant NSCLC after failure of prior standard therapy. The specifics of the incidence, nature and severity data can be found under the Adverse Events section.
Time Frame: 31 months
Measure: Number; unit: participants
Arm/Group | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD | RMC-4630 200 mg BIW D1D2 + Sotorasib 960 mg QD
Number analyzed (Participants) | 4 | 43
participants
  Serious Adverse Events | 3 | 43
  Other (Not Including Serious) Adverse Events | 4 | 43

ADVERSE EVENTS:
Time Frame: 1. RMC-4630 140 mg + Sotorasib 960 mg QD *Up to 31 months 2. RMC-4630 200 mg D1D2 + Sotorasib 960 mg QD *Up to 31 months
Description: Subjects were counted once within each system organ class and preferred term. Percentages were based on the number of all treated subjects in each column.
Arm/Group | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD | RMC-4630 200 mg BIW D1D2 + Sotorasib 960 mg QD
All-Cause Mortality (participants affected / at risk) | 3/4 | 21/43
Serious Adverse Events (participants affected / at risk) | 3/4 | 43/43
Other Adverse Events (participants affected / at risk) | 4/4 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD (N=4) | RMC-4630 200 mg BIW D1D2 + Sotorasib 960 mg QD (N=43)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Catheter site pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Perforated ulcer (General disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 4
Diverticulitis (Infections and infestations) | 0 | 2
Bacterial sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RMC-4630 140 mg BIW D1D2 + Sotorasib 960 mg QD (N=4) | RMC-4630 200 mg BIW D1D2 + Sotorasib 960 mg QD (N=43)
Anaemia (Blood and lymphatic system disorders) | 0 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 27
Nausea (Gastrointestinal disorders) | 3 | 8
Vomiting (Gastrointestinal disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 3
Oedema peripheral (General disorders) | 2 | 11
Fatigue (General disorders) | 2 | 7
Pyrexia (General disorders) | 0 | 6
Influenza like illness (General disorders) | 0 | 4
Face oedema (General disorders) | 0 | 3
Asthenia (General disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 3
Pneumonia (Infections and infestations) | 1 | 6
Bronchitis (Infections and infestations) | 0 | 5
COVID-19 (Infections and infestations) | 0 | 5
Bacteraemia (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 20
Aspartate aminotransferase increased (Investigations) | 3 | 19
Blood alkaline phosphatase increased (Investigations) | 2 | 14
Gamma-glutamyltransferase increased (Investigations) | 1 | 12
Blood bilirubin increased (Investigations) | 0 | 5
Lipase increased (Investigations) | 0 | 4
Blood creatine phosphokinase increased (Investigations) | 0 | 3
Blood creatinine increased (Investigations) | 0 | 3
C-reactive protein increased (Investigations) | 0 | 3
Platelet count decreased (Investigations) | 0 | 3
Weight decreased (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 8
Dehydration (Metabolism and nutrition disorders) | 1 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Dizziness (Nervous system disorders) | 0 | 4
Headache (Nervous system disorders) | 0 | 4
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications by investigators must be reviewed and approved by the sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT05054725/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT05054725/SAP_001.pdf